CLINICAL TRIAL: NCT00003241
Title: Phase II Study of Phenylacetate in Pediatric Patients With Central Nervous System Tumors
Brief Title: Phenylacetate in Treating Children With Recurrent or Progressive Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Texas Children's Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: TCCC-H-5057; CDR0000066116 (Registry Identifier: PDQ (Physician Data Query)); NCI-98-C-0107D; NCI-T96-0070
Record Dates: First submitted 1999-11-01; First posted 2004-09-10 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2000-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent childhood brain tumor; childhood high-grade cerebral astrocytoma; untreated childhood brain stem glioma; recurrent childhood brain stem glioma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood medulloblastoma; recurrent childhood ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Medulloblastoma; Familial ependymoma | interventions — phenylacetic acid

INTERVENTIONS:
Drug: phenylacetate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of phenylacetate in treating children with recurrent or progressive brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of phenylacetate in terms of response rate and time to progression in children with recurrent or progressive brain tumors, or with previously untreated poor prognosis brain tumors. II. Assess the toxicity of phenylacetate in these patients treated at the maximum tolerated dose. III. Determine the correlation between serum steady state phenylacetate levels and toxicity or response in these patients.

OUTLINE: Patients are stratified by histologic type (anaplastic astrocytoma and glioblastoma multiforme vs brain stem glioma vs medulloblastoma and primitive neuroectodermal tumors vs ependymoma vs low grade glioma vs others). Patients receive phenylacetate as a continuous intravenous infusion on days 1-28. Courses of treatment are given continuously without rest. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients are followed weekly.

PROJECTED ACCRUAL: A total of 9-30 patients per stratum will be accrued for this study in 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent or progressive brain tumors including the following: Anaplastic astrocytoma and glioblastoma multiforme Brain stem glioma Medulloblastoma or primitive neuroectodermal tumors present in supratentorial or posterior fossa locations Ependymoma Low grade gliomas Other Measurable or evaluable disease by CT or MRI OR Histologically confirmed previously untreated glial tumors including: Brain stem glioma Glioblastoma multiforme Measurable disease after surgery

PATIENT CHARACTERISTICS: Age: 2 to 21 Performance status: Karnofsky 50-100% (over 10 years of age) Lansky 50-100% (under 10 years of age) Life expectancy: At least 8 weeks Hematopoietic: Absolute neutrophil count greater than 1,000/mm3 Platelet count greater than 50,000/mm3 Hemoglobin greater than 7.0 g/dL Transfusion support allowed after bone marrow transplantation or extensive radiation Hepatic: Bilirubin less than 1.5 mg/dL SGPT less than 2 times normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance greater than 60 mL/min Other: Not pregnant or nursing Fertile patients must use effective contraception during and for 6 months after study No significant systemic illness including infections No amino acidurias or organic acidemias

PRIOR CONCURRENT THERAPY: Biologic therapy: Recovered from all prior immunotherapy No concurrent prophylactic hematopoietic growth factors Chemotherapy: At least 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosourea) and recovered No other concurrent cancer chemotherapy Endocrine therapy: Stable or decreasing dosage of dexamethasone for intracranial pressure within 2 weeks of study entry No concurrent dexamethasone used as an antiemetic Radiotherapy: At least 8 weeks since prior radiotherapy to evaluable lesions and recovered Surgery: At least 4 months since prior radiosurgery Other: No other concurrent investigational agents

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1998-05; Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Bomgaars, MD, Study Chair — Texas Children's Cancer Center
Locations (6):
- United States (6):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Pediatric Oncology Branch, Bethesda, Maryland
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Texas Children's Cancer Center, Houston, Texas